CLINICAL TRIAL: NCT05295602
Title: The Relationship of Radiological Lower Limb Alignment and Grade of the Knee Osteoarthritis With the Position of the Tibial Tuberosity
Brief Title: The Influence of Coronally Knee Alignment on the Tibial Tuberosity Rotation
Status: Completed | Type: Observational
Sponsor: Valdoltra Orthopedic Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Valdoltra - TT rotation
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee alignment; knee arthroplasty; tibial component rotation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group: A CT scan of both legs will be made in patient scheduled for a primary knee arthroplasty. No other additional intervention will be made apart from those already routinely used for the operation.
  Interventions: Radiation: CT scan

INTERVENTIONS:
Radiation: CT scan — CT of lower leg

SUMMARY:
The primary aim of this study is to find a possible correlation between tibial tuberosity rotation and coronal leg alignment. If correlation exists, a more individual tibial component rotation might be proposed during a total knee arthroplasty.

DETAILED DESCRIPTION:
A malalignment of the tibial component is a possible source of pain after a total knee arthroplasty. Currently, an internal rotation of the tibial component of 18 degrees is considered as a golden standard. The value was obtained as an average rotation in the osteoarthritic knees scheduled for a total knee arthroplasty.

It is known that the femur internally rotates with the increasing valgus alignment. It would seem logical that also tibial rotation correlates with the coronal limb alignment (varus-valgus). The plan is to measure the native tibial rotation (angle between the transposed epicondylar line and the posterior cruciate-tibial tuberosity line). In order to get the necessary accuracy a CT of lower legs will be obtained in patients waiting for the knee replacement. If there is a correlation between the angles the adjustment of the tibial component rotation more to the patient's anatomy could be proposed.

A secondary outcome measure is the possible correlation between the proximal femoral anteversion and the tibial tuberosity rotation. The hypothesis is that the extensor mechanism follows the proximal femoral orientation. With increasing femoral anteversion (increases with valgus angle) the femoral part of the knee rotates internally. In order to keep the extensor mechanism in the direction of walking, a more lateralized position of the tibial tuberosity is expected.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring knee arthroplasty

Exclusion Criteria:

* women in reproductive age, patients with leg deformities and previous hip/knee surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients waiting for the knee arthroplasty will be asked to participate. Patients with pre-existing deformities will not be enrolled. Additionally, women in reproductive age will also not be enrolled to avoid unnecessary radiation risks.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Correlation between coronal alignment and tibial tuberosity rotation | Before surgery
  A hip-knee-ankle angle and a tibial rotation angle (angle between the transposed epicondylar line) will be calculated from the CT scan of the leg. A correlation between both angles will be analysed using the Spearmans's coefficient.

SECONDARY OUTCOMES:
Correlation between femoral anteversion and tibial tuberosity position | Before surgery
  A femoral anteversion angle (angle between femoral hip neck and posterior condylar knee line) and tibial tuberosity position (angle between posterior condylar line and posterior cruciate - tibial tuberosity line) will be measured and examined for correlation using a Spearman's coefficient.
Difference in tibial tuberosity position according to the osteoarthritis grade | Before surgery
  Tibial tuberosity position will be compared according to the Kellgren-Lawrence grade with the ANOVA

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Strahovnik, Principal Investigator — Valdoltra Orthopaedic Hospital
Locations (1):
- Orthopaedic Hospital Valdoltra, Ankaran, Slovenia

IPD SHARING:
Plan to Share IPD: No